CLINICAL TRIAL: NCT05944770
Title: ASPIRE (Advancing Science Partnerships for Indoor Reductions of Smoke Exposures)-Health Tulare County
Brief Title: ASPIRE Health Tulare County
Acronym: ASPIREHealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Ann Chelminski, Principal Investigator, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-0965
Record Dates: First submitted 2023-05-31; First posted 2023-07-13 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Tract Diseases; Cardiovascular Diseases
Keywords: air pollution; wildfire smoke; wildland fire smoke; air filtration; indoor air quality
MeSH Terms: conditions — Respiratory Tract Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention or control group.
Who Masked: Participant
Masking Description: The control air filtration device will have a filter that looks like the intervention filter but is much less effective. A cover "shroud" will be placed over the air filtration device so that differences in components will not be noticeable to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Subjects in the treatment arm will use a DIY portable air cleaner made by attaching a highly effective furnace filter (MERV 13) and carbon absorbent to a box fan.
  Interventions: Other: DIY portable air cleaner with a highly effective filter
- Control arm (Sham Comparator): Subjects in the control arm will use a DIY portable air cleaner with a sham filter. All subjects will receive education on air quality, wildfire smoke, and health.
  Interventions: Other: DIY portable air cleaner with sham filtration

INTERVENTIONS:
Other: DIY portable air cleaner with a highly effective filter — A portable air filtration device that can be homemade ("DIY"), constructed by attaching a highly effective air filter (MERV13 rating or higher) to a 20 inch box fan to filter air pollutants including particulate matter of size 2.5 micrometers diameter or greater.
  Arms: Intervention arm
Other: DIY portable air cleaner with sham filtration — A portable air filtration device that can be homemade ("DIY") by attaching an air filter to a 20 inch box fan. The portable air cleaner with sham filtration with have a filter that is not effective for filtration of fine particulate matter, including that in wildfire smoke.
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to compare indoor air quality and health in people exposed to air pollution, including possible exposure to wildfire smoke. The study will test the effect of using a do-it-yourself (DIY) air cleaner when air pollution is present to answer the following questions:

* Do health outcomes differ between participants who use a DIY PAC and those who use a sham air cleaner?
* How effective is the DIY air cleaner in reducing indoor concentrations of fine particles (PM2.5), and volatile organic compounds found in wildfire smoke? OR How effective is the DIY air cleaner in reducing indoor concentrations of fine and coarse particles (i.e., PM 10)?
* What are barriers to use of a DIY air cleaner and what factors facilitate its use?

Participants will be asked to do the following:

* Participate in 5 home visits from study staff between July - October 2023
* Have an air quality sensor placed in the participant's bedroom for the whole study period
* Have a small sensor attached to the main door of the participant's house to record when the door is open or closed (important for air quality inside)
* Allow researchers to take air and dust samples in the participant's bedroom
* Run a DIY air cleaner in the participant's bedroom for at least 6 nights while the participant sleeps
* Complete 2 interviews
* Allow study staff to collect 3 fingerstick blood samples
* Allow study staff to collect 3 samples of fluid from inside the nose
* Use the study air cleaner in the participant's bedroom during the study period

The investigators will measure air quality in participating homes and measure health outcomes for participants. The investigators will compare outcomes of participants who use a DIY air cleaner with filters that work well to those of participants who use a DIY air cleaner with a placebo filter (one that does not work well to remove the air pollutants of concern). The goal of the study is to see if using the effective air cleaner leads to better health outcomes and indoor air quality.

DETAILED DESCRIPTION:
Background and rationale: The motivation for this research is that wildfires have been increasing in frequency and severity in recent years. Wildfire smoke is associated with numerous adverse health outcomes. Public health guidance during wildfire events has included recommendations to stay indoors, close doors and windows, and use portable air cleaners (PACs) to clean the smoke that infiltrates the indoor environment. Studies support the effectiveness of PACs in reducing indoor fine particulate matter, (PM2.5=fine particles 2.5 micrometers in diameter or smaller), one of the main components of concern in wildfire smoke.

Evidence of whether PAC use is associated with health benefits is mixed. In addition, commercially-available PACs can be expensive and hard to access. An affordable alternative that gained attention during the COVID-19 pandemic is a Do-It-Yourself (DIY) PAC, made from a box fan and high efficiency filter(s). Laboratory studies have shown DIY PACs to have excellent clean air delivery rates (CADR, a measure of effectiveness) with respect to fine particulate matter. However, their evidence in real-world settings is limited. Researchers have acknowledged that behaviors, such as turning on/off the fans, could have major impacts on efficacy.

The current study aims to examine the effect of PACs on indoor air quality and health during wildfire smoke exposure. The investigators will conduct this research in an agricultural community in central California that has experienced wildfire smoke exposure and routinely experiences dust. According to local partners, most residents of this county do not already own PACs. One risk of planning a Randomized Control Trial (RCT) of wildfire smoke exposure is that wildfire smoke will not occur. For this reason, the investigators selected a community with historically elevated levels of particle pollution (PM2.5, PM10, dust) in the fall and winter months as the study site. If wildfire smoke exposure does not occur during the study period, the efficacy of the DIY PACs on indoor air quality and health will be tested during periods of dust/high particle pollution exposure (anticipated October 2023).

Up to 120 recruited and consented study participants will be randomly divided into 2 groups. One group will use an effective DIY air cleaner (intervention); the other group will use a sham DIY air cleaner (control). All groups will have the same basic exposure to ambient air pollution.

Qualified participants will agree to have air quality sensors and door monitors placed in their home (bedroom and main exterior door). Air quality will be measured continuously during the study period. Other study activities will occur intermittently, during 5 visits by study staff to the participant's home. These activities will include completing 2 symptom and demographic questionnaires, collecting air and dust samples from inside the homes and collecting biological samples at 3 visits (capillary blood (by fingerstick) and nasal epithelial lining fluid). Blood and nasal fluid collected will be assessed for markers of inflammation and immune system activation. The investigators hypothesize that subjects in the intervention group will have reduced concentrations of measured air pollutants in their indoor air samples and lower levels of markers of inflammation compared to those in the control group. The investigators further hypothesize that symptoms, particularly related to respiratory inflammation, will differ between intervention (air filtration) and control (sham filtration) groups. Baseline measurements and post-intervention period measurements will be compared for intra-individual change and differences between study groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Has access to telephone and/or the internet for study communication
* Is a resident of Tulare County, California
* Is proficient in English or Spanish for study communication

Exclusion Criteria:

* Anyone in the household smokes (tobacco, vape, or other) inside the home
* Plans to move before November 2023
* Regularly travels or sleeps away from home (e.g., once a week or more)
* Already owns and uses a portable air cleaner
* Lives in a multi-unit home with a shared central HVAC system
* Has a bleeding disorder, such as hemophilia (taking a blood thinning medication does not exclude)
* Takes any of the following anti-inflammatory medications regularly: abatacept (Orencia), adalimumab(Humira), anakinra (Kineret), anifrolumab (Saphnelo), apremilast (Otezla), azathioprine (Imuran),certolizumab pegol (Cimzia), etanercept (Enbrel), golimumab (Simponi Aria), hydroxychloroquine(Plaquenil), infliximab (Remicade), ixekizumab (Taltz), leflunomide (Arava), methotrexate(Rheumatrex, Trexall), prednisone (Deltasone), sulfasalazine (Azulfidine), rituximab (Rituxan,MabThera), sarilumab (Kevzara), tocilizumab (Actemra)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change in concentrations of biomarkers of inflammation between treatment and control groups | Measured at baseline (pre-intervention) and at two timepoints, at least 3 days apart, during the portable air cleaner usage period (intervention)
  Markers of inflammation include C-reactive protein obtained from fingerstick blood samples

SECONDARY OUTCOMES:
Difference in change in concentrations of biomarkers of inflammation between treatment and control groups | Measured at Baseline and at two timepoints, at least 3 days apart, during the portable air cleaner usage period (intervention)
  Markers of inflammation obtained from nasal epithelial lining fluid analyses
Symptom data | At baseline and at one timepoint during portable air cleaner use
  Symptom/clinical data obtained from questionnaires

OTHER OUTCOMES:
air quality measurements | Continuous measurement lasting up to 15 weeks
  Concentrations of PM2.5, PM10 and volatile organic compounds in air inside participants' homes

CONTACTS AND LOCATIONS:
Overall Officials: Ann N Chelminski, MD, MPH, Principal Investigator — Environmental Protection Agency (EPA); Nayamin Martinez, MPH, Principal Investigator — Central California Environmental Justice Network
Locations (1):
- Central California Environmental Justice Network, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cascio WE. Wildland fire smoke and human health. Sci Total Environ. 2018 May 15;624:586-595. doi: 10.1016/j.scitotenv.2017.12.086. Epub 2017 Dec 27. PMID 29272827
- [Background] 2. U.S. Environmental Protection Agency. Create a Clean Room to Protect Indoor Air Quality During a Wildfire. 2022; https://www.epa.gov/indoor-air-quality-iaq/create-clean-room-protect-indoor-air-quality-during-wildfire. Accessed September 30, 2022.
- [Background] Cheek E, Guercio V, Shrubsole C, Dimitroulopoulou S. Portable air purification: Review of impacts on indoor air quality and health. Sci Total Environ. 2021 Apr 20;766:142585. doi: 10.1016/j.scitotenv.2020.142585. Epub 2020 Sep 30. PMID 33121763
- [Background] 4. Program CTAQ. Box fan filter, a DIY users guide. 2022; https://www.cct-enr.com/box-fan-filter. Accessed September 16, 2022.
- [Background] 5. Puget Sound Clean Air Agency. DIY Air Filter. https://pscleanair.gov/525/DIY-Air-Filter. Accessed September 16, 2022.
- [Background] Srikrishna D. Can 10x cheaper, lower-efficiency particulate air filters and box fans complement High-Efficiency Particulate Air (HEPA) purifiers to help control the COVID-19 pandemic? Sci Total Environ. 2022 Sep 10;838(Pt 1):155884. doi: 10.1016/j.scitotenv.2022.155884. Epub 2022 May 14. PMID 35580674
- [Background] Holder AL, Halliday HS, Virtaranta L. Impact of do-it-yourself air cleaner design on the reduction of simulated wildfire smoke in a controlled chamber environment. Indoor Air. 2022 Nov;32(11):e13163. doi: 10.1111/ina.13163. PMID 36437679
- [Background] Batterman S, Du L, Mentz G, Mukherjee B, Parker E, Godwin C, Chin JY, O'Toole A, Robins T, Rowe Z, Lewis T. Particulate matter concentrations in residences: an intervention study evaluating stand-alone filters and air conditioners. Indoor Air. 2012 Jun;22(3):235-52. doi: 10.1111/j.1600-0668.2011.00761.x. Epub 2012 Feb 4. PMID 22145709
- See also: Create a clean room to protect indoor air quality during a wildfire — https://www.epa.gov/indoor-air-quality-iaq/create-clean-room-protect-indoor-air-quality-during-wildfire